CLINICAL TRIAL: NCT03748758
Title: Evaluation of Safety of Repeated Doses of OP0201 Metered Dose Inhaler Compared to Placebo in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novus Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: OP0201-C-002
Record Dates: First submitted 2018-11-13; First posted 2018-11-21 (Actual); Results first posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Healthy Adult Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Drug: OP0201 (30 mg) (Active Comparator): Cohort A- 30 mg per day X 14 days
  Interventions: Combination Product: Drug: OP0201
- Drug: Placebo (Placebo Comparator): Cohort A- 0 mg per day X 14 days Cohort B- 0 mg per day X 14 days
  Interventions: Combination Product: Drug: Placebo
- Drug: OP0201 (60 mg) (Active Comparator): Cohort B-60 mg per day X 14 days
  Interventions: Combination Product: Drug: OP0201

INTERVENTIONS:
Combination Product: Drug: OP0201 — Drug OP0201
  Arms: Drug: OP0201 (30 mg); Drug: OP0201 (60 mg)
Combination Product: Drug: Placebo — Placebo
  Arms: Drug: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of two dose levels of OP0201 and placebo, when administered intranasally in healthy adults subjects.

ELIGIBILITY:
Inclusion Criteria includes but is not limited to:

1. Body mass index of 18 to 30 kg/m2 (inclusive) and a minimum body weight of 50 kg at Screening.
2. Able and willing to follow study instructions (including compliance with daily study treatment administration) and likely to complete all required study visits as assessed by the Investigator's judgement.
3. Female subjects must agree to use an acceptable method of contraception (for pregnancy considerations and contraceptive requirements).
4. Female subjects who are of childbearing potential must have a negative urine pregnancy test result at Screening and Day -1 prior to randomization.
5. Male subjects must agree to use contraception
6. Subjects must agree to refrain from immersing their head fully under water (eg, swimming, diving) from the time of signed informed consent until after the study exit visit.
7. Physiologic tympanogram classified as Type A (normal) by the Investigator or designee.

Exclusion Criteria includes but is not limited to:

1. History or presence of significant medical condition or a clinically significant abnormal finding, as determined by the Investigator.
2. Presence of a clinically significant abnormal olfactory test finding at Screening defined as a total UPSIT score <35 (for females) and <34 (for males).
3. Clinically significant ear disorder/disease currently or within 6 weeks prior to Screening.
4. History of tympanostomy tubes in one or both ears within 1 year prior to Screening.
5. Upper respiratory tract infection or pharyngitis currently or within 6 weeks prior to Screening.
6. Allergy or sinus conditions (eg, sinusitis, non-specific nasal inflammation) currently or within 6 weeks prior to Screening.
7. Clinically relevant blockage of one or both nasal passages, in the Investigator's opinion.
8. Gastroesophageal reflux disease currently or within 6 weeks prior to Screening.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vince and Associates, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://novustherapeutics.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Drug: OP0201 Cohort A 30 mg Per Day: Cohort A- 30 mg per day X 14 days
  Drug: OP0201: Drug OP0201
- Drug: OP0201 Cohort B 60 mg Per Day: Cohort B-60 mg per day X 14 days
  Drug: OP0201: Drug OP0201
- Drug: Placebo: 0 mg per day X 14 days
  Drug: Placebo: Placebo
Period: Overall Study
Arm/Group | Drug: OP0201 Cohort A 30 mg Per Day | Drug: OP0201 Cohort B 60 mg Per Day | Drug: Placebo
Started | 12 | 12 | 6
Completed | 12 | 12 | 5
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug: OP0201 Cohort A 30 mg Per Day | Drug: OP0201 Cohort B 60 mg Per Day | Drug: Placebo | Total
Number analyzed (Participants) | 12 | 12 | 6 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (7.2) | 32.2 (6.2) | 35.3 (10.4) | 33.5 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 4 | 12
  Male | 6 | 10 | 2 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 8 | 3 | 16
  White | 7 | 4 | 3 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 6 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With of Adverse Events
Time Frame: 21 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Drug: OP0201 Cohort A 30 mg Per Day | Drug: OP0201 Cohort B 60 mg Per Day | Drug: Placebo
Number analyzed (Participants) | 12 | 12 | 6
Participants | 5 | 9 | 4

2. Secondary Outcome: Evaluation of Systemic Exposure of DPPC: Observed DPPC Serum Concentration (µg/mL) by Nominal Timepoint
Description: This will be evaluated by collecting blood on Day 1 baseline, Day 14 at 30 minutes pre-dose, and 5, 20, 35, and 50 minutes post-dose only in OP0201 Cohort B 60 mg per day
Time Frame: Day 1 and Day 14
Population: It is pre-specified to collect and report data for only "Cohort B" and "Placebo" Arms/Groups per protocol. The Number of participants analyzed for Cohort B at Day 14, 30 mins pre-dose and 5 mins post-dose is one less compared to other timepoints due to exclusion of serum samples that had missing collection times.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Drug: OP0201 Cohort B 60 mg Per Day/ Day 1 Baseline; Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 30 Mins Predose; Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 5 Mins; Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 20 Mins; Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 35 Mins; Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 50 Mins: Cohort B-60 mg per day X 14 days Drug: OP0201: Drug OP0201
- Drug: Placebo/ Day 1 Baseline; Drug: Placebo/ Day 14: 30 Mins Predose; Drug: Placebo/ Day 14: 5 Mins; Drug: Placebo/ Day 14: 20 Mins; Drug: Placebo/ Day 14: 35 Mins; Drug: Placebo/ Day 14: 50 Mins: 0 mg per day X 14 days Drug: Placebo: Placebo
Arm/Group | Drug: OP0201 Cohort B 60 mg Per Day/ Day 1 Baseline | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 30 Mins Predose | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 5 Mins | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 20 Mins | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 35 Mins | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 50 Mins | Drug: Placebo/ Day 1 Baseline | Drug: Placebo/ Day 14: 30 Mins Predose | Drug: Placebo/ Day 14: 5 Mins | Drug: Placebo/ Day 14: 20 Mins | Drug: Placebo/ Day 14: 35 Mins | Drug: Placebo/ Day 14: 50 Mins
Number analyzed (Participants) | 12 | 11 | 11 | 12 | 12 | 12 | 2 | 2 | 2 | 2 | 2 | 2
µg/mL | 10.05 (2.585) | 10.18 (2.703) | 10.35 (2.832) | 9.954 (2.475) | 9.813 (2.368) | 10.04 (2.564) | 9.525 (2.652) | 12.86 (6.145) | 14.03 (7.319) | 13.20 (6.505) | 12.80 (6.930) | 13.39 (6.668)

3. Secondary Outcome: Evaluation of Systemic Exposure of CP: Observed CP Serum Concentrations (µM) by Nominal Timepoint
Description: as for outcome 2
Time Frame: Day 1 and Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Drug: OP0201 Cohort B 60 mg Per Day/ Day 1 Baseline | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 30 Mins Predose | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 5 Mins | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 20 Mins | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 35 Mins | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 50 Mins | Drug: Placebo/ Day 1 Baseline | Drug: Placebo/ Day 14: 30 Mins Predose | Drug: Placebo/ Day 14: 5 Mins | Drug: Placebo/ Day 14: 20 Mins | Drug: Placebo/ Day 14: 35 Mins | Drug: Placebo/ Day 14: 50 Mins
Number analyzed (Participants) | 12 | 11 | 11 | 12 | 12 | 12 | 2 | 2 | 2 | 2 | 2 | 2
µM | 299.503 (61.999) | 290.103 (35.978) | 293.473 (56.417) | 279.852 (44.170) | 279.289 (44.424) | 276.788 (45.493) | 298.519 (126.157) | 363.530 (178.783) | 387.945 (200.583) | 363.476 (165.774) | 366.353 (195.732) | 368.159 (178.270)

4. Secondary Outcome: Evaluation of Systemic Exposure of DPPC: Baseline-corrected DPPC Serum Concentration (µg/mL) by Nominal Timepoint
Description: as for outcome 2
Time Frame: Day 1 and Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 30 Mins Predose | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 5 Mins | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 20 Mins | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 35 Mins | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 50 Mins | Drug: Placebo/ Day 14: 30 Mins Predose | Drug: Placebo/ Day 14: 5 Mins | Drug: Placebo/ Day 14: 20 Mins | Drug: Placebo/ Day 14: 35 Mins | Drug: Placebo/ Day 14: 50 Mins
Number analyzed (Participants) | 11 | 11 | 12 | 12 | 12 | 2 | 2 | 2 | 2 | 2
µg/mL | 0.309 (0.347) | 0.871 (0.787) | 0.383 (0.453) | 0.300 (0.407) | 0.447 (0.446) | 3.333 (3.490) | 4.505 (4.660) | 3.678 (3.850) | 3.278 (4.274) | 3.865 (4.009)

5. Secondary Outcome: Evaluation of Systemic Exposure of CP: Baseline-corrected CP Serum Concentrations (µM) by Nominal Timepoint
Description: as for outcome 2
Time Frame: Day 1 and Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 30 Mins Predose | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 5 Mins | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 20 Mins | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 35 Mins | Drug: OP0201 Cohort B 60 mg Per Day/ Day 14: 50 Mins | Drug: Placebo/ Day 14: 30 Mins Predose | Drug: Placebo/ Day 14: 5 Mins | Drug: Placebo/ Day 14: 20 Mins | Drug: Placebo/ Day 14: 35 Mins | Drug: Placebo/ Day 14: 50 Mins
Number analyzed (Participants) | 11 | 11 | 12 | 12 | 12 | 2 | 2 | 2 | 2 | 2
µM | 8.341 (15.478) | 15.625 (18.781) | 6.697 (14.869) | 6.818 (13.839) | 5.699 (10.410) | 65.011 (52.626) | 89.426 (74.425) | 64.957 (39.617) | 67.834 (69.575) | 69.641 (52.113)

ADVERSE EVENTS:
Time Frame: End of study (Day 21)
Arm/Group | Drug: OP0201 Cohort A 30 mg Per Day | Drug: OP0201 Cohort B 60 mg Per Day | Drug: Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 5/12 | 9/12 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drug: OP0201 Cohort A 30 mg Per Day (N=12) | Drug: OP0201 Cohort B 60 mg Per Day (N=12) | Drug: Placebo (N=6)
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Feeling cold (General disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Olfactory test abnormal (Investigations) | 0 | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No information, data or results shall be used by the Institution, Investigator or any other individual or entity other than the Sponsor. The use of Study Results by any party other than Sponsor requires prior written approval by the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT03748758/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT03748758/SAP_001.pdf